CLINICAL TRIAL: NCT02633280
Title: A Predictive "Molecular Biology Signature" for Diagnosis and Treatment of Chronic Obstructive Pulmonary Disease
Brief Title: Biomarkers for Diagnosis and Treatment of COPD
Acronym: BmiRCOPD
Status: Completed | Type: Observational
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Luca Gallelli, MD, University of Catanzaro
Other Study IDs: COPD
Record Dates: First submitted 2015-11-27; First posted 2015-12-17 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- COPD-Untreated (Group 1): In this Group will be enrolled patients of both sex and older than 40-years with COPD stage GOLD 2 and 3 that did not receive COPD treatment in the last 6 months (beta 2 agonists, corticosteroids, anticholinergics).
- COPD-uncontrolled (Group 2): In this Group will be enrolled patients of both sex and older than 40-years with COPD stage GOLD 2 and 3 that receive a COPD treatment (e.g. beta 2 agonists, corticosteroids, anticholinergics) but with a post-bronchodilator FEV1< 80% and an FEV1/FVC < 0.7 or with 1-2 exacerbation/year
- Control subjects (Group 3): In this Group will be enrolled patients of both sex and older than 40 years; (2) will be free from lung disease as determined by a physician; (3) will have a normal spirometry (FEV1> 85% and FEV1/FVC > 0.7)

SUMMARY:
COPD is an inflammatory disease characterized by enhanced chronic airway and lung inflammatory responses to noxious agents (e.g. smoke, pollutants) and progressive airflow limitation. In COPD patients there is a spillover of peripheral lung inflammation into systemic circulation resulting in increased level of various inflammatory markers such as: IL-1β, IL-6, IL-8, and TNF-α.

Diagnosis, now, is based on clinical evaluation and spirometry test and COPD treatment includes the use of LABA, LAMA and corticosteroids.

To data no plasmatic marker able to identify the stage of COPD and the response to the treatment have been documented . The aim of this study is to evaluate in COPD patients the role of microRNA as predictive biomarker, of the disease in order to have a signature of miRs typically of COPD

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a heterogeneous respiratory disorder affecting more than 200 million patients worldwide. It is characterized by enhanced chronic airway and lung inflammatory responses to noxious agents (e.g. smoke, pollutants) and progressive airflow limitation.

Both, prevalence and incidence of this disease are continuously increasing, thus the investigators can predict that in 2020 it will be the third important cause of death in the world.

Several immune system cells (e.g. macrophages, eosinophils) and biochemical mediators (e.g. tumor necrosis factor-alpha, transforming growth factor beta, Interleukins and metalloproteases) are involved in its development and in symptom severity.

It has been suggested that in COPD patients there is a spillover of peripheral lung inflammation into systemic circulation resulting in increased level of various inflammatory markers such as: IL-1β, IL-6, IL-8, and TNF-α. Those biomolecules are responsible of various complication associated with COPD such as cardiovascular disease, hypertension and skeletal muscle weakness to name a few. It is worth to note that the increase of systemic inflammatory markers is also responsible of diabetes, obesity and metabolic syndrome development in COPD patients.

Diagnosis, now, is based on clinical evaluation and spirometry test and COPD treatment includes the use of LABA, LAMA and corticosteroids. Therefore, an early diagnosis in order to asses a specific treatment it is mandatory.

Sarioglu et al.,reported that systemic inflammatory markers levels (in plasma) TNFα, IL-6 and C-reactive protein, persist in the stable period in 110 COPD patients and the C-reactive protein levels correlate with the COPD Assessment Test.

However, C-reactive protein is not a specific marker, while to date more appropriate marker(s) could be represented by microRNA (miR) a key class of gene expression regulators, emerging as crucial players in various biological processes such as cellular proliferation and differentiation, development and apoptosis.

In this concern, Stolzenburg et al., documented, in an experimental model of COPD, that miR-1343 reduces the expression of both isoform of TGF-b receptor 1 and 2, directly targeting their 3' UTRs mRNA region, suggesting a role in the improvement of lung fibrosis.

To date, no other data have been performed yet on this topic. In the present project the investigators would like to screen with nCounter GX Human Inflammation Kit a comprehensive number of 249 human genes known to be differentially expressed in inflammation. The gene list represents a broad range of inflammation-related pathways. In parallel miRs screening will be performed (800 in a single reaction tube) using NanoString Technology Platform. This technology is robust and sensitive and today is used for the validation of New Generation Sequence (NGS) data. Our aim is to evaluate in COPD patients the role of miRs as predictive biomarker, of the disease in order to have a signature of miRs typically of COPD. The signature could be used to monitoring the therapeutic application of drugs used in COPD as well as to asses a Prediction COPD Diagnostic test.

The absence of a plasmatic marker able to identify the stage of disease and the response to the treatment leads to COPD exacerbation and progression, this represent, in the real life, a common problem during COPD treatment and is also related with an increase of sanitary health costs. Last year, the European health bill for COPD treatment increased by USD 10 million and the market is thought to increase up to USD 37.7 million by 2030.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosed according to the GOLD criteria

Exclusion Criteria:

* allergy to corticosteroids or to bronchodilators
* neurodegenerative diseases
* autoimmune diseases
* inability to use inhalers
* progressive serious medical conditions (such as cancer, AIDS or end-stage renal disease)
* infectious diseases

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: An open label, parallel groups study, will be performed after it is approve by the Ethical committee and before the beginning of the study, all participants will be informed about the aim, procedures, risks and benefits of the study and they will provide a written informed consent
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2016-04; Primary Completion 2017-04 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Change of miR expression at 6 and 12 months | 6 and 12 months
  Change of miR expression in COPD-groups (Groups 1 and 2 ) vs control-Group

SECONDARY OUTCOMES:
correlation between miRs expression and clinical outcome | 6 and 12 months
  correlation between miRs and clinical outcome evaluated through the COPD Assessment Test (CAT) and the modified Medical Research Council (mMRC) dispnea scale
correlation between miRs expression and the development of adverse drug reaction | 6 and 12 months
  correlation between miRs and clinical outcome evaluated through the Naranjo probability scale
correlation between miRs expression and inflammatory markers | 6 and 12 months
  correlation between miRs expression and plasma levels of ILs, TNF-Alpha, C reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Luca Gallelli, MD, Principal Investigator — University of Catanzaro
Locations (3):
- Italy (3):
  - UCCP, Badolato, Catanzaro
  - UCCP, Borgia, Catanzaro
  - UCCP, Catanzaro

REFERENCES:
- [Result] Garvey C. Recent updates in chronic obstructive pulmonary disease. Postgrad Med. 2016;128(2):231-8. doi: 10.1080/00325481.2016.1118352. Epub 2015 Dec 1. PMID 26560514
- [Result] Vestbo J, Hurd SS, Agusti AG, Jones PW, Vogelmeier C, Anzueto A, Barnes PJ, Fabbri LM, Martinez FJ, Nishimura M, Stockley RA, Sin DD, Rodriguez-Roisin R. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2013 Feb 15;187(4):347-65. doi: 10.1164/rccm.201204-0596PP. Epub 2012 Aug 9. PMID 22878278
- [Result] Barnes PJ. Chronic obstructive pulmonary disease: effects beyond the lungs. PLoS Med. 2010 Mar 16;7(3):e1000220. doi: 10.1371/journal.pmed.1000220. PMID 20305715
- [Result] Sarioglu N, Hismiogullari AA, Bilen C, Erel F. Is the COPD assessment test (CAT) effective in demonstrating the systemic inflammation and other components in COPD? Rev Port Pneumol (2006). 2016 Jan-Feb;22(1):11-7. doi: 10.1016/j.rppnen.2015.08.007. Epub 2015 Oct 31. PMID 26534740
- [Result] Stolzenburg LR, Wachtel S, Dang H, Harris A. miR-1343 attenuates pathways of fibrosis by targeting the TGF-beta receptors. Biochem J. 2016 Feb 1;473(3):245-56. doi: 10.1042/BJ20150821. Epub 2015 Nov 5. PMID 26542979
- [Result] Watt J, Ganapathi P. COPD: Novel therapeutics and management strategies--SMi's 7th Annual Conference (October 19-20, 2015--London, UK). Drugs Today (Barc). 2015 Oct;51(10):613-7. doi: 10.1358/dot.2015.51.10.2409817. PMID 26583304
- [Result] Agusti A, Edwards LD, Rennard SI, MacNee W, Tal-Singer R, Miller BE, Vestbo J, Lomas DA, Calverley PM, Wouters E, Crim C, Yates JC, Silverman EK, Coxson HO, Bakke P, Mayer RJ, Celli B; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) Investigators. Persistent systemic inflammation is associated with poor clinical outcomes in COPD: a novel phenotype. PLoS One. 2012;7(5):e37483. doi: 10.1371/journal.pone.0037483. Epub 2012 May 18. PMID 22624038